CLINICAL TRIAL: NCT03411044
Title: Fitmore Hip Stem Post-Market Clinical Follow-Up (PMCF) Study
Brief Title: Fitmore Hip Stem PMCF Study: A Multi-centre, Non-comparative, Prospective Post-market Clinical Follow-up Study.
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 09H06
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Prosthesis Failure
Keywords: Total Hip Arthroplasty; Fitmore; Minimal Invasive Surgery; Short Stem
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with a Fitmore Hip Stem: Subjects in need of a total hip arthroplasty who met the inclusion/exclusion criteria and who received the Fitmore Hip Stem.
  Interventions: Device: Fitmore Hip Stem

INTERVENTIONS:
Device: Fitmore Hip Stem

SUMMARY:
A multi-centre, non-comparative, prospective post-market clinical follow-up study to obtain survival, clinical and radiographic outcomes data on the Zimmer Fitmore Hip Stem.

DETAILED DESCRIPTION:
The objective of this post market surveillance study is to obtain outcome data on the Fitmore Hip Stem by analysis of standard scoring systems, radiographs and adverse event records, and thus to assess the long-term performance and safety of this implant.

The Fitmore Hip Stem is a short and curved uncemented stem that allows preservation of the greater trochanter and of the gluteal muscles.

Indication/Target Population: Patients suffering from severe hip pain and disability requiring total hip arthroplasty.

Study Design: A multi-centre, non-comparative, prospective post-marketing study.

Targeted Number of Subjects: 500. Data Collection: Collection of preoperative, intra-operative and immediate post-operative data; follow-up visits at 6-12 weeks, 1, 2, 3, 5, 7 and 10 years post-operatively.

Recruitment period: 24 months. Clinical Assessments: Evaluations will be made using the Harris Hip Score, the Oxford Hip Score, the SF-12 Physical and Mental Health summary measures, the EQ-5D (EuroQol) and radiographically.

Safety Assessments: Safety will be assessed by appropriate recording and reporting of adverse events throughout the study. The Fitmore Hip Stem is CE marked, commercially available and has been pre-clinically tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are capable of understanding the doctor"s explanations, following his instructions and who are able to participate in the follow-up program.
* Patients who have given written consent to take part in the study by signing the "Patient Consent Form".
* 18 years minimum.
* Male and female.
* Patients suffering from severe hip pain and disability requiring hip surgery or as indicated in the treatment of a fracture.

Exclusion Criteria:

* Patients who are unwilling or unable to give consent or to comply with the follow-up program.
* Pregnancy.
* Patients who are skeletally immature.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe hip pain and disability requiring hip surgery using the Fitmore Hip Stem, who meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2008-02-08 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (5):
- Germany (2):
  - Auguste Viktoria Klinik, Bad Oeynhausen
  - Universitätsklinikum Carl Gustav Carus, Dresden
- Clinica San Michele, Albenga, Italy
- Kantonsspital Graubünden, Chur, Switzerland
- The Yorkshire Clinic, Bingley, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Suffering From Severe Hip Pain and Disability Requiring Total Hip Arthroplasty.: Subjects in need of THA who met the inclusion/exclusion criteria and who received the Fitmore Stem
Period: Overall Study
Arm/Group | Patients Suffering From Severe Hip Pain and Disability Requiring Total Hip Arthroplasty.
Started | 420
Completed | 230
Not Completed | 190
Not completed — Death | 30
Not completed — Withdrawal by Subject | 48
Not completed — Lost to Follow-up | 78
Not completed — Adverse Event | 30
Not completed — Missing status | 4

BASELINE CHARACTERISTICS:
Population: Patients suffering from severe hip pain and disability requiring hip surgery or as indicated in the treatment of a fracture.
Groups:
- Patients Suffering From Severe Hip Pain and Disability Requiring Total Hip Arthroplasty.: Patients suffering from severe hip pain and disability requiring hip surgery or as indicated in the treatment of a fracture.
Arm/Group | Patients Suffering From Severe Hip Pain and Disability Requiring Total Hip Arthroplasty.
Number analyzed (Participants) | 420
Age, Categorical [Count of Participants; unit: Participants]
  Study Population: <=18 years | 0
  Study Population: Between 18 and 65 years | 420
  Study Population: >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 230
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 70
  United Kingdom | 80
  Switzerland | 123
  Germany | 147

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score
Description: The Harris hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care Professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). The total score can vary from a range of 0 - 100. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70.
Time Frame: Preop, 6 - 12 weeks, 1 year, 2 year, 3 year, 5 year, 7 and 10 years
Population: Study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 358
score on a scale
  Preop | 50.0 (17.1)
  6 - 12 weeks | 80.6 (14.8)
  1 Year | 94.5 (8.0)
  2 Year | 94.5 (9.5)
  3 Year | 94.2 (10.0)
  5 Year | 93.5 (11.3)
  7 Year | 93.6 (11.2)
  10 Year | 92.6 (12.1)

2. Primary Outcome: Radiographic Evaluations
Description: Radiographic evaluation was assessed at the time points listed below in order to identify potential adverse events.
Time Frame: 6 - 12 weeks and 7 years
Population: The significant radiographic findings reported for all patients during the course of the study is presented in the results section below for all follow up time points of occurrence.
Measure: Number; unit: participants
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 164
participants
  6 - 12 weeks | 2
  7 Year | 1

3. Primary Outcome: Survivorship
Description: The primary endpoint for this study is implant survival at 10 years which is assessed by revision of the Fitmore Hip Stem calculated using the Kaplan-Meier Survival Estimation. The survivorship with Kaplan-Meier (K-M) was calculated at 10 year for endpoint revision of any component.
Time Frame: 10 years post surgery
Population: All study patients involved in the study.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 420
percentage | 96.85 [94.14 to 98.32]

4. Secondary Outcome: EQ5D
Description: The EuroQol 5 Dimension (EQ-5D) is a standardized Instrument widely used to measure health status. It is a self reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, selfcare, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. The EQ-5D-5L score ranges from -0.59 to 1, where 1 is the best possible health state. The Visual Analogue Scale (VAS) is a vertical scale ranges from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her self-rated health.
Time Frame: Preop, 6-12 weeks, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year and 10 Year
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 314
score on a scale
  Preop EQ-5D-5L | 0.4 (0.3)
  6 - 12 Weeks EQ-5D-5L: number analyzed (Participants) | 260
  6 - 12 Weeks EQ-5D-5L | 0.8 (0.2)
  1 Year EQ-5D-5L: number analyzed (Participants) | 219
  1 Year EQ-5D-5L | 0.9 (0.2)
  2 Year EQ-5D-5L: number analyzed (Participants) | 221
  2 Year EQ-5D-5L | 0.9 (0.2)
  3 Year EQ-5D-5L | 0.9 (0.2)
  5 Year EQ-5D-5L: number analyzed (Participants) | 226
  5 Year EQ-5D-5L | 0.9 (02)
  7 Year EQ-5D-5L: number analyzed (Participants) | 267
  7 Year EQ-5D-5L | 0.9 (0.2)
  10 Year EQ-5D-5L: number analyzed (Participants) | 221
  10 Year EQ-5D-5L | 0.9 (0.2)
  Preop VAS: number analyzed (Participants) | 250
  Preop VAS | 60.0 (19.0)
  6 - 12 Weeks VAS: number analyzed (Participants) | 259
  6 - 12 Weeks VAS | 74.5 (14.6)
  1 Year VAS: number analyzed (Participants) | 218
  1 Year VAS | 80.2 (14.3)
  2 Year VAS: number analyzed (Participants) | 211
  2 Year VAS | 79.1 (16.6)
  3 Year VAS: number analyzed (Participants) | 303
  3 Year VAS | 80.4 (15.3)
  5 Year VAS: number analyzed (Participants) | 233
  5 Year VAS | 80.2 (15.0)
  7 Year VAS: number analyzed (Participants) | 245
  7 Year VAS | 79.0 (16.2)
  10 Year VAS: number analyzed (Participants) | 220
  10 Year VAS | 78.1 (16.3)

5. Secondary Outcome: SF-12 Physical and Mental Functional Scores
Description: The SF-12 is a multipurpose short-form (SF) generic measure of health status. It consists of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Scores ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: Preop, 6-12 Weeks, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year and 10 Year
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 297
score on a scale
  Preop SF-12 physical: number analyzed (Participants) | 209
  Preop SF-12 physical | 27.1 (9.6)
  6-12 Weeks SF-12 physical: number analyzed (Participants) | 198
  6-12 Weeks SF-12 physical | 39.1 (9.5)
  1 Year SF-12 physical: number analyzed (Participants) | 162
  1 Year SF-12 physical | 49.5 (8.6)
  2 Year SF-12 physical: number analyzed (Participants) | 185
  2 Year SF-12 physical | 50.0 (9.1)
  3 Year SF-12 physical | 48.9 (9.2)
  5 Year SF-12 physical: number analyzed (Participants) | 208
  5 Year SF-12 physical | 50.3 (8.7)
  7 Year SF-12 physical: number analyzed (Participants) | 236
  7 Year SF-12 physical | 49.2 (9.3)
  10 Year SF-12 physical: number analyzed (Participants) | 201
  10 Year SF-12 physical | 47.4 (10.5)
  Preop SF-12 Mental: number analyzed (Participants) | 206
  Preop SF-12 Mental | 54.2 (9.6)
  6-12 Weeks SF-12 Mental: number analyzed (Participants) | 202
  6-12 Weeks SF-12 Mental | 56.6 (8.1)
  1 Year SF-12 Mental: number analyzed (Participants) | 170
  1 Year SF-12 Mental | 54.7 (7.3)
  2 Year SF-12 Mental: number analyzed (Participants) | 195
  2 Year SF-12 Mental | 55.1 (7.7)
  3 Year SF-12 Mental: number analyzed (Participants) | 293
  3 Year SF-12 Mental | 53.7 (8.2)
  5 Year SF-12 Mental: number analyzed (Participants) | 217
  5 Year SF-12 Mental | 53.0 (8.1)
  7 Year SF-12 Mental: number analyzed (Participants) | 244
  7 Year SF-12 Mental | 54.2 (8.7)
  10 Year SF-12 Mental: number analyzed (Participants) | 212
  10 Year SF-12 Mental | 54.2 (7.0)

6. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (warst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The Score ranges from 0 - 100 and the outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27.
Time Frame: Preop, 6-12 Weeks, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year and 10 Year
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With a Fitmore Hip Stem
Number analyzed (Participants) | 329
score on a scale
  Preop: number analyzed (Participants) | 308
  Preop | 19.3 (8.1)
  6-12 Weeks: number analyzed (Participants) | 256
  6-12 Weeks | 36.2 (7.5)
  1 Year: number analyzed (Participants) | 212
  1 Year | 42.8 (7.4)
  2 Year: number analyzed (Participants) | 232
  2 Year | 43.5 (6.8)
  3 Year | 43.3 (6.8)
  5 Year: number analyzed (Participants) | 235
  5 Year | 43.0 (7.5)
  7 Year: number analyzed (Participants) | 269
  7 Year | 44.2 (6.4)
  10 Year: number analyzed (Participants) | 218
  10 Year | 43.7 (6.3)

ADVERSE EVENTS:
Time Frame: Operative, 6-12 weeks, 1, 2, 3, 5, 7, 10 years
Arm/Group | Subjects With a Fitmore Hip Stem
All-Cause Mortality (participants affected / at risk) | 30/420
Serious Adverse Events (participants affected / at risk) | 40/420
Other Adverse Events (participants affected / at risk) | 132/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With a Fitmore Hip Stem (N=420)
Femoral Pain (Musculoskeletal and connective tissue disorders) | 9 — The section shows the hip related Adverse Events
Infection (Musculoskeletal and connective tissue disorders) | 8 — Deep Infection <6 Weeks Infection, systemic sepsis Superficial Infection
Other Hip Related Complication (Musculoskeletal and connective tissue disorders) | 6
Deep Vein Thrombosis (Musculoskeletal and connective tissue disorders) | 3
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 4
Hematoma (Musculoskeletal and connective tissue disorders) | 3
Femoral Implant Loosening (Musculoskeletal and connective tissue disorders) | 2
Fracture of Femoral Shaft (Musculoskeletal and connective tissue disorders) | 2
Fracture of Femoral Neck (Musculoskeletal and connective tissue disorders) | 2
Fracture of Trochanter (Musculoskeletal and connective tissue disorders) | 2
Nerve Deficit (Musculoskeletal and connective tissue disorders) | 1
Other General Complication (Musculoskeletal and connective tissue disorders) | 2 — Remaining drainage with THA
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With a Fitmore Hip Stem (N=420)
Other General Complication (Musculoskeletal and connective tissue disorders) | 19 — Coxathrosis, Depression, Dementia, Adipositas, Angiomyolipoma,
Other General Complication (Musculoskeletal and connective tissue disorders) | 19 — Contralateral Hip or Knee
Other Hip Related Complication (General disorders) | 19 — Cancer, Gastritis, Blood pressure,Scoliosis, Hernia, Back pain, Stent Implantation, Shingles.
Other General Complications (General disorders) | 19 — Arthrosis, Pain, Osteoathritis,
Other General Complications (General disorders) | 19 — Ankle Athrosis, Asthma, Diabetes.
Other General Complications (General disorders) | 19 — Bronchitis, Stenosis, Shoulder problems.
Other General Complication (General disorders) | 18 — Gastritis, Hernia, Back pain, Shingles, Asthma.

LIMITATIONS AND CAVEATS:
Due to the COVID 19 pandemic, many study patients could not return for the 10 year follow up resulting to drop out. In addition, one study site which enrolled 80 cases could not continue to follow the study patients at the 7 year follow up due to lack of resources to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-11-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03411044/Prot_SAP_000.pdf